CLINICAL TRIAL: NCT03819075
Title: An Evaluation Of Effectiveness Of A Combined Er:YAG And Nd:YAG Laser Protocol For Treatment Of Peri-Implantitis: A Randomized Controlled Trial
Brief Title: Combined Er:YAG And Nd:YAG Laser Protocol For Treatment Of Peri-Implantitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luis Monteiro (Other)
Responsible Party: Sponsor-Investigator, Luis Monteiro, DMD, Phd, Auxiliar Professor at the IUCS in Periodontal Surgical Clinic, Oral Pathology and Biopathology, Cooperativa de Ensino Superior, Politécnico e Universitário
Organization: Cooperativa de Ensino Superior, Politécnico e Universitário (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26/CE-IUCS/2018
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Peri-Implantitis
Keywords: laser; Er:YAG; Nd:YAG; periimplantitis; randomized controlled trial
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Two groups; laser and control
Who Masked: Outcomes Assessor
Masking Description: Clinical measurements will be performed by an evaluator unaware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): For the laser group we will use a Lightwalker Laser (Fotona) with a Er:YAG 2940 nm and Nd:YAG 1064 nm wavelengths units.
  Interventions: Device: Lightwalker Laser (Fotona)
- Control (Active Comparator): Standard periimplantitis treatment will be conducted in the control group.
  Interventions: Other: standard

INTERVENTIONS:
Device: Lightwalker Laser (Fotona) — For the laser group we will use a Lightwalker Laser (Fotona) with a Er:YAG 2940 nm and Nd:YAG 1064 nm wavelengths units. The laser protocol will follow the instructions of the manufacturer (TwinLight protocol) and consists of degranulation of necrotic soft tissue and bone, implant surface disinfection and creating spot bleeding in bone with Er:YAG and deep disinfection and biomodulation with Nd:YAG.
  Other Names: TwinLight periimplantitis
  Arms: Laser
Other: standard — Granulation tissue elimination, mechanical instrumentation of the implant surface and curettage of intraosseous or supracrestally bone defects will be accomplished using plastic curets, under irrigation with sterile saline solution. Cotton pellets soaked in sterile saline solution will be use to clean debris and remains of removed tissue.
  Arms: Control

SUMMARY:
A laser treatment for periimplantitis using two different wavelengths (Er:YAG and Nd:YAG) will be compared to standard treatment in a randomized clinical trial.

DETAILED DESCRIPTION:
The general aim of this study is to evaluate the clinical outcome of the treatment of peri-implantitis using a combination of a Er:YAG and Nd:YAG laser protocol or using a conventional mechanical treatment in patients with a diagnosis of peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

* at least one implant with peri-implantitis
* no serious mobility of the implants
* written informed consent of the voluntary participant in the study
* availability of participant for control visits for a follow-up of at least 12 months without interruptions

Exclusion Criteria:

* serious systematic disease
* pregnancy
* current use of photosensitive drugs, bisphosphonate medication or antibiotics
* patients who do not want to follow post treatment recommendation of oral hygiene and follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2018-03-03 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment success | 6 months
  Treatment success defined as implant survival with the absence of peri-implant probing depths (PD) greater than 5 mm with concomitant bleeding/suppuration and absence of progression of peri-implant bone loss.

SECONDARY OUTCOMES:
Plaque index | 1 month
  (PI)
Plaque index | 3 months
  (PI)
Plaque index | 6 months
  (PI)
Plaque index | 12 months
  (PI)
Bleeding on probing | 1 month
  (BOP) evaluated as present if bleeding was evident within 30 s after probing, or absent, if no bleeding was noticed within 30 s after probing.
Bleeding on probing | 3 months
  evaluated as present if bleeding was evident within 30 s after probing, or absent, if no bleeding was noticed within 30 s after probing.
Bleeding on probing | 6 months
  evaluated as present if bleeding was evident within 30 s after probing, or absent, if no bleeding was noticed within 30 s after probing.
Bleeding on probing | 12 months
  evaluated as present if bleeding was evident within 30 s after probing, or absent, if no bleeding was noticed within 30 s after probing.
Probing depth | 1 month
  measured from the mucosal margin to the bottom of the pocket.
Probing depth | 3 months
  measured from the mucosal margin to the bottom of the pocket.
Probing depth | 6 months
  measured from the mucosal margin to the bottom of the pocket.
Probing depth | 12 months
  measured from the mucosal margin to the bottom of the pocket.
Mucosal recession | 1 month
  measured from the mucosal margin to the bottom of the pocket.
Mucosal recession | 3 months
  measured from the mucosal margin to the bottom of the pocket.
Mucosal recession | 6 months
  measured from the mucosal margin to the bottom of the pocket.
Mucosal recession | 12 months
  measured from the mucosal margin to the bottom of the pocket.
Clinical attachment level gain | 1 month
  Difference in clinical attachment level at baseline and follow up.
Clinical attachment level gain | 3 months
  Difference in clinical attachment level at baseline and follow up.
Clinical attachment level gain | 6 months
  Difference in clinical attachment level at baseline and follow up.
Clinical attachment level gain | 12 months
  Difference in clinical attachment level at baseline and follow up.
Quality of life questionnaire | 0 months
  Oral Health Impact Profile-14 on the scale from 0 to 56 with higher scores indicating a poorer oral health-related quality of life.
Quality of life questionnaire | 1 month
  Oral Health Impact Profile-14 on the scale from 0 to 56 with higher scores indicating a poorer oral health-related quality of life.
Quality of life questionnaire | 3 months
  Oral Health Impact Profile-14 on the scale from 0 to 56 with higher scores indicating a poorer oral health-related quality of life.
Quality of life questionnaire | 6 months
  Oral Health Impact Profile-14 on the scale from 0 to 56 with higher scores indicating a poorer oral health-related quality of life.
Quality of life questionnaire | 12 months
  Oral Health Impact Profile-14 on the scale from 0 to 56 with higher scores indicating a poorer oral health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Monteiro, DMD, PhD, Principal Investigator — Instituto Universitário de Ciências da Saude, CESPU
Locations (1):
- Instituto Universitário de Ciências da Saude, CESPU, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No